CLINICAL TRIAL: NCT06759337
Title: The Effect of Stress Ball Used During Intra Uterine Insemination on Pain, Anxiety, Comfort and Physiological Parameters: A Randomized Controlled Study
Brief Title: The Effect of Stress Ball Used During Intra Uterine Insemination on Pain, Anxiety, Comfort and Physiological Parameters
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Emine Özge AVCI, mSc, nurse, TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2024/148; Erciyes University (Other: Erciyes University)
Record Dates: First submitted 2024-12-28; First posted 2025-01-06 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2024-12

CONDITIONS: Infertility Assisted Reproductive Technology; Infertility, Female
Keywords: Assisted Reproductive Techniques; Stress Ball; Pain; Anxiety; Comfort; Physiological Parameters; infertility
MeSH Terms: conditions — Infertility, Female; Pain; Anxiety Disorders; Infertility

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Stress Ball Group (Experimental): Participants are given a colored silicone stress ball (5-7 cm diameter) 5 minutes before the procedure. During the procedure, they are instructed to squeeze the ball twice after counting to 10 and repeat this until the procedure is complete.
  Interventions: Behavioral: Stress Ball Group
- Hand Holding/ Therapeutic Touch Group (Experimental): The researcher holds one of the participant's hands during catheter insertion and removal. The researcher's fingers are closed but not interlocked and placed gently on the participant's hand without additional movements or gloves.
  Interventions: Behavioral: Hand-Holding Group
- Control Group (No Intervention): Participants receive no additional intervention beyond the standard routine procedures.

INTERVENTIONS:
Behavioral: Stress Ball Group — Participants are given a colored silicone stress ball (5-7 cm diameter) 5 minutes before the procedure. During the procedure, they are instructed to squeeze the ball twice after counting to 10 and repeat this until the procedure is complete.
  Arms: Stress Ball Group
Behavioral: Hand-Holding Group — The researcher holds one of the participant's hands during catheter insertion and removal. The researcher's fingers are closed but not interlocked and placed gently on the participant's hand without additional movements or gloves.
  Arms: Hand Holding/ Therapeutic Touch Group

SUMMARY:
This study aimed to determine the effects of holding the patient's hand and using a stress ball during the Intrauterine Insemination procedure on pain, anxiety, comfort, and physiological parameters. This study will be conducted as a randomized controlled trial with a pre-test-post-test procedure in the IVF Unit of a Medical Faculty Hospital in Turkey. The study sample was planned to include 120 participants, 40 women each in the stress ball, hand-holding, and control groups. Data will be collected using the Personal Information Form, Visual Analog Scale, State Anxiety Inventory, and General Comfort Scale Short Form. In the Stress Ball Group, participants are given a colored silicone stress ball (5-7 cm diameter) 5 minutes before the procedure. During the procedure, they are instructed to squeeze the ball twice after counting to 10 and repeat this until the procedure is complete. In the Hand-Holding Group, the researcher holds one of the participant's hands during catheter insertion and removal. The researcher's fingers are closed but not interlocked and placed gently on the participant's hand without additional movements or gloves. In the Control Group, Participants receive no additional intervention beyond the standard routine procedures.

DETAILED DESCRIPTION:
Infertility is a significant social and health issue, negatively affecting couples, particularly women's biological, physical, and psychosocial well-being. Assisted reproductive techniques are utilized to help couples with infertility achieve parenthood (Taşkın, 2023). Among these techniques, the Intrauterine Insemination (IUI) procedure can lead to pain, anxiety, discomfort, and trauma, both from the procedure itself and from the emotional impact of infertility. Pain associated with trauma and anxiety may trigger adverse effects, such as increased catecholamine levels, reduced heart rate, blood pressure, and lung vital capacity, due to the activation of the sympathetic nervous system (Yıldız Fındık and Soydaş Yeşilyurt, 2017; Vaajoki et al., 2012).

To alleviate acute pain and enhance comfort during IUI procedures, in addition to medical interventions, non-pharmacological methods with minimal side effects are also critical (Stewart and Cox-Davenport, 2015). One such approach is the attention distribution method, which enables brain receptors to shift focus away from painful stimuli, thereby reducing pain perception and improving control (Elmali and Balcı Akpinar, 2017). The use of stress balls as a non-pharmacological method of attention distribution is particularly noteworthy. Stress balls are accessible, cost-effective, and safe. Furthermore, their use offers a holistic approach, incorporating touch, healing, and therapeutic effects (Yanes et al., 2018). A review of the literature reveals various findings on the psychometric and vital sign changes-such as anxiety, stress, comfort, and compliance-associated with stress ball use during medical procedures, including colonoscopy, endoscopy, extracorporeal shock wave lithotripsy (ESWL), prostate biopsy, radiography, hemodialysis, intravenous (IV) procedures, and polymerase chain reaction (PCR) testing (Apaydin Cirik et al., 2023; Çakır and Evirgen, 2023; Özen et al., 2023; Karataş and Gezginci, 2023, 2022; Gezginci et al., 2018a; Karataş and Gezginci, 2018; Quan et al., 2016). Additionally, some studies highlight the therapeutic or healing benefits of touch in children and intensive care settings (Garrett and Riou, 2021). However, the specific effects of hand-holding and stress ball use on pain, anxiety, comfort, and physiological parameters during the IUI procedure have not yet been thoroughly investigated.

ELIGIBILITY:
Inclusion Criteria:

Intervention Group 1 (Stress Ball Group)

1. Agreeing to participate in the study with verbal and written consent,
2. Being between the ages of 18-50,
3. Being able to read and write in Turkish,
4. Not having a muscle or joint problem that prevents squeezing the stress ball
5. Having Intrauterine Insemination (insemination) as an infertility treatment,

Intervention Group 2 (Hand Holding Group)

1. Agreeing to participate in the study with verbal and written consent,
2. Being between the ages of 18-50,
3. Being able to read and write in Turkish,
4. Not having a problem with holding hands
5. Having Intrauterine Insemination (insemination) as an infertility treatment,

Control Group

1. Agreeing to participate in the study with verbal and written consent,
2. Being between the ages of 18-50,
3. Being able to read and write in Turkish,
4. Having Intrauterine Insemination (insemination) as an infertility treatment, To have an insemination (vaccination) procedure,

Exclusion Criteria:

Intervention Group (Stress Ball Group)

1. Use any analgesic agent at least 24 hours before the procedure,
2. Having a chronic pain disorder,
3. Abandoning the completion of the data collection forms,
4. Needing urgent intervention by a physician during or immediately after the procedure,
5. Having any psychiatric disease,
6. Having a visual, hearing, speech, physical or mental disability,
7. Wanting to leave the study at any stage,
8. Not applying the stress ball application as requested

Intervention Group (Hand Holding Group)

1. Use any analgesic agent at least 24 hours before the procedure,
2. Having a chronic pain disorder,
3. Being uncomfortable with the hand-holding application,
4. Abandoning the completion of the data collection forms,
5. Needing urgent intervention by a physician during or immediately after the procedure,
6. Having any psychiatric disease,
7. Having visual, hearing, speech, having a physical or mental disability,
8. Wanting to leave the study at any stage,

Control Group

1. Use any analgesic agent at least 24 hours before the procedure,
2. Having a chronic pain disorder,
3. Stopping the completion of the data collection forms,
4. Needing urgent intervention by a physician during or immediately after the procedure,
5. Having any psychiatric disease,
6. Having a visual, hearing, speech, physical or mental disability,
7. Wanting to leave the study at any stage,

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 120 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Personal Information Form | The researcher will apply 10 minutes before the IUI procedure and 15 minutes after the procedure to women who are kept under observation in the patient monitoring room after the IUI procedure.
  This form, which includes the characteristics of the patients, consists of 10 questions, including age, education level, marital status, employment status, income level, type of infertility, duration of infertility problem, and cause of infertility. The patient's physiological parameters (pulse, respiration, systolic blood pressure (SBP), diastolic blood pressure (DBP), and oxygen saturation values (SpO2) before and after the procedure will also be recorded using this form.
Visual Analog Scale | The researcher will apply 10 minutes before the IUI procedure and 15 minutes after the procedure to women who are kept under observation in the patient monitoring room after the IUI procedure.
  It will be used to determine the pain intensity experienced by infertile women during IUI. The pain level varies between 0-10, and the increase in the marked numerical value indicates an increase in the pain level. In the VAS evaluation, 0=no pain, 1-4=mild pain, 5-6=moderate pain, and 7-10=severe pain (Zielinski et al., 2020).
State Anxiety Inventory | The researcher will apply 10 minutes before the IUI procedure and 15 minutes after the procedure to women who are kept under observation in the patient monitoring room after the IUI procedure.
  The scale Spielberger et al. (1970) developed to measure the individual's state and trait anxiety level, reliability, and validity in Turkish was conducted by Öner and Le Compte (1983). The scale measures anxiety. It consists of two sub-units that are measured separately: state anxiety requires the individual to describe how they feel at a certain moment and under certain conditions, and trait anxiety requires the individual to describe how they generally feel. In this study, the state anxiety scale will be used since the anxiety that the individual feels indirectly from the stressful situation they are in will be evaluated. The total score obtained from the scale varies between 20 and 80, with a high score indicating a high level of anxiety.
General Comfort Scale Short Form | The researcher will apply 10 minutes before the IUI procedure and 15 minutes after the procedure to women who are kept under observation in the patient monitoring room after the IUI procedure.
  The Kolcaba (2006) scale was developed to measure patients' comfort. The scale consists of 28 items in 6-point Likert type in 3 sub-dimensions: relief (9), relaxation (9), and overcoming problems sub-dimension (10 items). The highest total score from the scale is 168 points; the lowest total score is 28 points (Çıtlık et al., 2018)

CONTACTS AND LOCATIONS:
Overall Officials: Hümeyra TÜLEK DENİZ, MSc, Principal Investigator — Kafkas University
Locations (1):
- Erciyes University Medical Faculty Hospital IVF Unit, Kayseri, Melikgazi, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
There has been no planning on this matter.

REFERENCES:
- [Background] Apaydin Cirik V, Turkmen AS, Ayaz M. Effectiveness of stress ball and relaxation exercises on polymerase chain reaction (RRT-PCR) test-induced fear and pain in adolescents in Turkiye. J Pediatr Nurs. 2023 Jul-Aug;71:135-140. doi: 10.1016/j.pedn.2022.12.001. Epub 2022 Dec 14. PMID 36526480
- [Background] Cakir SK, Evirgen S. Three Distraction Methods for Pain Reduction During Colonoscopy: A Randomized Controlled Trial Evaluating the Effects on Pain and Anxiety. J Perianesth Nurs. 2023 Oct;38(5):e1-e7. doi: 10.1016/j.jopan.2023.02.007. Epub 2023 Aug 10. PMID 37565937
- [Background] Elmali H, Balci Akpinar R. The effect of watching funny and unfunny videos on post-surgical pain levels. Complement Ther Clin Pract. 2017 Feb;26:36-41. doi: 10.1016/j.ctcp.2016.11.003. Epub 2016 Nov 9. PMID 28107847
- [Background] Garrett B, Riou M. A rapid evidence assessment of recent therapeutic touch research. Nurs Open. 2021 Sep;8(5):2318-2330. doi: 10.1002/nop2.841. Epub 2021 Mar 20. PMID 33742792
- [Background] Genc H, Korkmaz M, Akkurt A. The Effect of Virtual Reality Glasses and Stress Balls on Pain and Vital Findings During Transrectal Prostate Biopsy: A Randomized Controlled Trial. J Perianesth Nurs. 2022 Jun;37(3):344-350. doi: 10.1016/j.jopan.2021.09.006. Epub 2022 Apr 7. PMID 35397973
- [Background] Gezginci E, Iyigun E, Kibar Y, Bedir S. Three Distraction Methods for Pain Reduction During Cystoscopy: A Randomized Controlled Trial Evaluating the Effects on Pain, Anxiety, and Satisfaction. J Endourol. 2018 Nov;32(11):1078-1084. doi: 10.1089/end.2018.0491. PMID 30280915
- [Background] Gezginci E, Iyigun E, Yalcin S, Bedir S, Ozgok IY. Comparison of Two Different Distraction Methods Affecting the Level of Pain and Anxiety during Extracorporeal Shock Wave Lithotripsy: A Randomized Controlled Trial. Pain Manag Nurs. 2018 Jun;19(3):295-302. doi: 10.1016/j.pmn.2017.09.005. Epub 2017 Dec 14. PMID 29248604
- [Background] Karatas TC, Gezginci E. The Effect of Using a Stress Ball During Endoscopy on Pain, Anxiety, and Satisfaction: A Randomized Controlled Trial. Gastroenterol Nurs. 2023 Jul-Aug 01;46(4):309-317. doi: 10.1097/SGA.0000000000000739. Epub 2023 May 17. PMID 37199436
- [Background] Ozen N, Berse S, Tosun B. Effects of using a stress ball on anxiety and depression in patients undergoing hemodialysis: A prospective, balanced, single-blind, crossover study. Hemodial Int. 2023 Oct;27(4):411-418. doi: 10.1111/hdi.13102. Epub 2023 Jun 15. PMID 37318078
- [Background] Sadeghi T, Mohammadi N, Shamshiri M, Bagherzadeh R, Hossinkhani N. Effect of distraction on children's pain during intravenous catheter insertion. J Spec Pediatr Nurs. 2013 Apr;18(2):109-14. doi: 10.1111/jspn.12018. Epub 2013 Mar 5. PMID 23560582
- [Background] Shekhar S, Suprabha BS, Shenoy R, Rao A, Rao A. Effect of active and passive distraction techniques while administering local anaesthesia on the dental anxiety, behaviour and pain levels of children: a randomised controlled trial. Eur Arch Paediatr Dent. 2022 Jun;23(3):417-427. doi: 10.1007/s40368-022-00698-7. Epub 2022 Mar 10. PMID 35274286
- [Background] Quan X, Joseph A, Nanda U, Moyano-Smith O, Kanakri S, Ancheta C, Loveless EA. Improving Pediatric Radiography Patient Stress, Mood, and Parental Satisfaction Through Positive Environmental Distractions: A Randomized Control Trial. J Pediatr Nurs. 2016 Jan-Feb;31(1):e11-22. doi: 10.1016/j.pedn.2015.08.004. Epub 2015 Sep 26. PMID 26395650
- [Background] Stewart M, Cox-Davenport RA. Comparative Analysis of Registered Nurses' and Nursing Students' Attitudes and Use of Nonpharmacologic Methods of Pain Management. Pain Manag Nurs. 2015 Aug;16(4):499-502. doi: 10.1016/j.pmn.2014.09.010. Epub 2014 Dec 12. PMID 25499026
- [Background] Vaajoki A, Pietila AM, Kankkunen P, Vehvilainen-Julkunen K. Effects of listening to music on pain intensity and pain distress after surgery: an intervention. J Clin Nurs. 2012 Mar;21(5-6):708-17. doi: 10.1111/j.1365-2702.2011.03829.x. Epub 2011 Aug 15. PMID 21843204
- [Background] Yanes AF, Weil A, Furlan KC, Poon E, Alam M. Effect of Stress Ball Use or Hand-holding on Anxiety During Skin Cancer Excision: A Randomized Clinical Trial. JAMA Dermatol. 2018 Sep 1;154(9):1045-1049. doi: 10.1001/jamadermatol.2018.1783. PMID 30027283
- [Background] Yilmaz D, Gunes UY. The effect on pain of three different nonpharmacological methods in peripheral intravenous catheterisation in adults. J Clin Nurs. 2018 Mar;27(5-6):1073-1080. doi: 10.1111/jocn.14133. Epub 2018 Jan 8. PMID 29076581
- [Background] Zielinski J, Morawska-Kochman M, Zatonski T. Pain assessment and management in children in the postoperative period: A review of the most commonly used postoperative pain assessment tools, new diagnostic methods and the latest guidelines for postoperative pain therapy in children. Adv Clin Exp Med. 2020 Mar;29(3):365-374. doi: 10.17219/acem/112600. PMID 32129952